CLINICAL TRIAL: NCT00527774
Title: Impact of Hepatitis C Virus Infection on Insulin Resistance and Inflammatory Biomarkers in Patients With Maintenance Hemodialysis
Brief Title: Effect of HCV Infection on Insulin Resistance and Malnutrition-inflammation Complex Syndrome in Regular Hemodialysis Patients
Status: Completed | Type: Observational
Sponsor: St. Martin De Porress Hospital (Other)
Collaborators: National Taiwan University (Other)
Responsible Party: Sponsor
Other Study IDs: P0702
Record Dates: First submitted 2007-09-10; First posted 2007-09-11 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-05

CONDITIONS: Hepatitis C; Hemodialysis; Quality of Life; Mortality; Hospitalization
Keywords: Hepatitis C; malnutrition-inflammation complex syndrome (MICS); dialysis; mortality; hospitalization; health-related quality of life (HRQOL); peripheral arterial occlusive disease (PAOD)
MeSH Terms: conditions — Hepatitis C; Peripheral Arterial Occlusive Disease 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Check HCV viral load and genotype in first month and sixth month
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- A: HCV(+) maintenance hemodialysis patients
- B: HCV(-) maintenance hemodialysis patients

SUMMARY:
The purpose of this study is to study whether hepatitis C virus (HCV)infected maintenance hemodialysis (MHD)patients have distinct metabolic, inflammatory and adipokine characteristics that can be linked to poor clinical outcome and to examine the hypothesis that HCV infected MHD patients with metabolic syndrome have higher risks for hospitalization, cardiovascular and all-cause mortality.

DETAILED DESCRIPTION:
Background: High prevalence of hepatitis C virus (HCV) infection is noticed in Yun-Lin, Chiayi area in Taiwan. Patients with maintenance hemodialysis (MHD) in this area have the highest risk for HCV infection. Understanding the natural history of HCV and its association with inflammation, nutrition and outcomes in dialysis patients may provide more information for anti-HCV management strategies in dialysis and other patient populations.

Objective: We hypothesize that HCV infected MHD patients have distinct metabolic, and inflammatory characteristics that can be linked to adverse conditions and increased higher morbidity and mortality.

Design: A cross-sectional study is conducted in one regional teaching hospital with its medical alliance dialysis clinics. A cohort of 200 MHD patients including 70 HCV subjects are recruited. Basic data and dialysis characteristics are collected. Metabolic syndrome (MS) is defined according to International Diabetes Federation (IDF) consensus 2005. Insulin resistance (IR) is defined by HOMA index. Comorbidity is rated by Charlson Comorbidity Score. Malnutrition-inflammation score (MIS) is used to rate the severity of malnutrition-inflammation complex syndrome (MICS). Nutritional and appetite status are evaluated by appetite and diet assessment tool (ADAT) and anthropometric evaluation. Inflammatory status is measured by biomarkers such as serum concentrations of C-reactive protein, tumor necrosis factor-α, interleukin-1β, interleukin-6, adiponectin, leptin and plasminogen activator inhibitor-1. Ankle-brachial index (ABI)test is used to predict the severity of peripheral arterial occlusive disease (PAOD). We use Beck's depression inventory to assess depression status and apply SF36, WHOQOL and EQ-5D questionnaires to assess health-related quality of life (HRQOL). Outcome evaluations are based on mortality and hospitalizations followed prospectively for up to 6 months.

ELIGIBILITY:
Inclusion Criteria:

* The main inclusion criteria were those outpatients who were undergoing MHD for at least 8 weeks, were 18 years or older, and who signed the written consent form.

Exclusion Criteria:

* Patients with a clinical or laboratory evidence of active infectious diseases in the last 1 month before inclusion in the study, or life expectancy of less than 6 months, for example, because of a metastatic malignancy or terminal HIV disease, were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A cross-sectional study was conducted in one regional teaching hospital (St. Martin De Porres Hospital) in Chiayi City in Taiwan and its medical alliance dialysis clinics during Sept. 2007 to March 2008.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2007-09; Primary Completion 2008-02 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chung-Jing Wang, M.D., Study Chair — St. Martin De Porres Hospital; Kuan-Yu Hung, M.D. & Ph.D., Principal Investigator — Nephrology Section, Department of Internal Medicine, National Taiwan University and College of Medicine; Pau-Chung Chen, M.D. & Ph.D., Study Director — Institute of Occupational Medicine and Industrial Hygiene, College of Public Health, National Taiwan University
Locations (1):
- Hemodialysis Center, St. Martin De Porres Hospital, Chiayi City, Taiwan